CLINICAL TRIAL: NCT02227511
Title: Prospective Randomized Trial of Fruits or Nuts Eaten Between Regular Meals in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, Professor, MD, Head of Internal Medicine, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014/170-31
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Subjects
Keywords: fruit, nuts, liver fat, insulin, glucose; Focus of the study is to compare the often given advice to eat fruit, containing large amount of glucose and fructose, with nuts that are more rich in fat.
MeSH Terms: conditions — Fatty Liver; Insulin Resistance | interventions — Fruit; Nuts; Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fruit (Active Comparator): Participants are given +7kCal/kg body weight of fruit to be eaten as snack in between regular meals
  Interventions: Dietary Supplement: Fruits
- nuts (Active Comparator): Participants are given +7kCal/kg body weight of nuts to be eaten as snack in between regular meals
  Interventions: Dietary Supplement: Nuts

INTERVENTIONS:
Dietary Supplement: Fruits — Randomization to extra fruit or nuts as snacks
  Arms: fruit
Dietary Supplement: Nuts
  Other Names: Randomization to extra fruit or nuts as snacks
  Arms: nuts

SUMMARY:
Recruitment of 28 subjects that will be randomized to consume fruit or nuts as snacks between regular meals for two months. Laboratory tests for cardiovascular risk factors, metabolic rate, liver steatosis and physical activity are investigated ahead of start of the study and at the end of the trial period och two months. Participants will be allowed to buy fruits or nuts on their own but to keep track (diaries) of the amount consumed. They will be reimbursed for the costs of the snacks.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* significant diseases that can affect outcomes, mental disorders that can affect participation.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
amount of fat in the liver by magnetic resonance imaging | two months
  exact measurement of fat in the liver by liver spectroscopy

SECONDARY OUTCOMES:
cardiovascular risk factors | two months
  Collection of markers for cardiovascular risk including glucose, insulin, lipoproteins etc. Analyses will be performed from blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Fredrik H Nystrom, Linköping, Sweden

REFERENCES:
- [Derived] Agebratt C, Strom E, Romu T, Dahlqvist-Leinhard O, Borga M, Leandersson P, Nystrom FH. A Randomized Study of the Effects of Additional Fruit and Nuts Consumption on Hepatic Fat Content, Cardiovascular Risk Factors and Basal Metabolic Rate. PLoS One. 2016 Jan 20;11(1):e0147149. doi: 10.1371/journal.pone.0147149. eCollection 2016. PMID 26788923